CLINICAL TRIAL: NCT02500524
Title: A Randomised, Controlled, Assessor-blind, Parallel Group Clinical Trial to Assess the Efficacy, Safety and Acceptability of a Surfactant Based Lotion and a Permethrin Creme Rinse in the Treatment of Head Lice
Brief Title: Cocamide DEA vs Permethrin for Head Lice
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Medical Entomology Centre (Industry)
Collaborators: PN Lee Statistics and Computing Ltd (Unknown); Riemann a/s (Unknown)
Responsible Party: Principal Investigator, Ian F Burgess, Director, Medical Entomology Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTRL01
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pediculosis Capitis; Head Louse Infestation
MeSH Terms: interventions — coconut diethanolamide; Permethrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10% Cocamide diethanolamine (Experimental): 10% Cocamide DEA aqueous lotion is applied directly to dry hair on a single occasion and is washed off with shampoo after 60 minutes.
  Interventions: Drug: Cocamide diethanolamine
- 1% permethrin creme rinse (Active Comparator): 1% permethrin creme rinse is applied to shampooed and towel dried hair on a single occasion and left in situ for 10 minutes, then rinsed off with clean water.
  Interventions: Drug: Permethrin

INTERVENTIONS:
Drug: Cocamide diethanolamine — Topical lotion
  Other Names: Lauramine diethanolamine
  Arms: 10% Cocamide diethanolamine
Drug: Permethrin — Topical creme rinse
  Arms: 1% permethrin creme rinse

SUMMARY:
To assess the efficacy and safety of 10% Cocamide DEA and Lyclear creme rinse (permethrin1%) in the eradication of head lice. To assess the ability of each product to kill all viable ova and to assess patient acceptability of the product in use.

DETAILED DESCRIPTION:
A formulation of cocamide diethanolamine (DEA) surfactant was previously reported as showing efficacy to eliminate head louse infestation. This study has been designed to test those data using a new formulation of 10% cocamide DEA in an aqueous basis in comparison with the standard of care product 1% permethrin creme rinse. It is believed that surfactants like cocamide DEA are capable of eliminating lice resistant to conventional insecticides.

A planned total of 120 patients who, following examination, are found to suffer from active head lice infestation will be recruited to the trial. The patient will be treated with the appropriate product according to the randomization code from a pre-prepared listing in balanced blocks of 12.

10% Cocamide DEA is applied directly to dry hair and is washed off with shampoo after 60 minutes. Permethrin 1% creme rinse is applied to shampooed and towel dried hair and left in situ for 10 minutes, then rinsed off with clean water. Treatments will be applied by experienced investigators throughout the study. Assessments will be made by other investigators unaware of the treatment regimen used.

After treatment (day 0), follow up assessments will be performed on days 4, 7,10 then again at day 14 after which they will leave the study. Any adverse events or side effects from the treatments will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 4 who are found to have a head lice infection.
* Patients who give written informed consent or, if the patient is under 16 years of age, whose guardian gives written informed consent to participate in the study.
* Available for the duration of study i.e. 15 days.

Exclusion Criteria:

* Patients with a known sensitivity to pyrethroid, organophosphate, and/or carbamate insecticides, sensitivity to chrysanthemums and/or known sensitivity to paraben preservatives.
* Patients who have been treated with other head lice products within the last 4 weeks.
* Patients who have undergone a course of antibiotic treatment within the last 4 weeks.
* Patients who have any persistent skin disorder of the scalp (i.e. eczema, chronic dermatitis, psoriasis).
* Patients with asthma
* Patients whose hair has been bleached, colour treated or permed within the last 4 weeks.
* Pregnant or nursing mothers.
* Patients who have participated in another clinical trial within 1 month prior to entry to this study.
* Patients who have already participated in this clinical trial.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 1998-07; Primary Completion 1999-01 (Actual); Study Completion 1999-01 (Actual)

PRIMARY OUTCOMES:
Elimination of infestation | 14 days
  No evidence of active head lice infestation 14 days after enrolment.

SECONDARY OUTCOMES:
The number of participants with treatment related adverse events as a measure of safety | 14 days
  No treatment related adverse events following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Burgess, Principal Investigator — Medical Entomology Centre
Locations (1):
- Medical Entomology Centre, Cambridge, United Kingdom